CLINICAL TRIAL: NCT00117637
Title: A Randomised, Open-label, Multi-centre Phase II Study of BAY43-9006 (Sorafenib) Versus Standard Treatment With Interferon Alpha-2a in Patients With Unresectable and/or Metastatic Renal Cell Carcinoma.
Brief Title: BAY43-9006 (Sorafenib) Versus Interferon Alpha-2a in Patients With Unresectable and/or Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11848; 2005-000544-86 (EudraCT Number)
Record Dates: First submitted 2005-06-30; First posted 2005-07-08 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal Cell Cancer; RCC; Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — Sorafenib; Interferons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- First Sorafenib (Nexavar, BAY43-9006) 400 mg then 600 mg (Experimental): Subjects received 2 tablets of Sorafenib (200 mg tablets) twice daily (bid) (ie 12-hourly) orally until progression (= first intervention period, 5.7 months [median] ) and 3 tablets of Sorafenib twice daily (ie 12-hourly) orally until the following progression (= second intervention period, 3.6 months [median]) on a continuous basis.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- First Interferon then Sorafenib (Nexavar, BAY43-9006) 400 mg (Active Comparator): Interferon (IFN) α-2a was administered at a dose of 9 million international units(MIU) subcutaneously three times a week until progression (= first intervention period, 5.6 months [median]). Subjects initially started with a single dose of 3 MIU IFN and increased the dose as rapidly as possible to 9 MIU IFN three times a week within 1 or 2 weeks in first intervention period.After first progression, subjects received 2 tablets of Sorafenib (200 mg tablets) twice daily (BID) (ie 12-hourly) until the next progression (=second intervention period, 5.3 months [median]).
  Interventions: Drug: Interferon

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Multi kinase inhibitor
  Arms: First Sorafenib (Nexavar, BAY43-9006) 400 mg then 600 mg
Drug: Interferon — Interferon
  Arms: First Interferon then Sorafenib (Nexavar, BAY43-9006) 400 mg

SUMMARY:
The purpose of the study is to:

* Find out if patients receiving BAY43-9006 will live longer without tumor progression than those receiving standard therapy with interferon alpha-2a
* Find out if a higher dose of BAY43-9006 can inhibit tumor progression in patients who progressed during standard dose treatment with BAY43-9006, and for how long these patients live without progression
* Find out how long patients live without progression who receive BAY43-9006 after failing to respond to standard therapy with interferon alpha-2a
* Find out in how many percent of patients BAY43-9006 prevents the growth of or shrinks kidney tumors and/or their metastases depending on treatment and dosage
* Find out if BAY43-9006 has any effect on the quality of life of patients with kidney cancer
* Find out the level of BAY43-9006 in the blood once per month and any changes in this level
* Find out whether BAY43-9006 effects are associated with specific biomarkers

DETAILED DESCRIPTION:
Analyses on Biomarkers were exploratory and assessed as tertiary objective of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time, without prejudice
* Male or female patients >= 18 years of age
* Patients who have a life expectancy of at least 12 weeks
* Patients, who suffer from unresectable and/or metastatic, measurable predominantly clear cell RCC (Renal Cell Carcinoma) histologically or cytologically documented
* Patients must have undergone prior (at the time of primary diagnosis) complete surgical excision of primary RCC tumor
* Patients must have had no prior systemic therapy for advanced RCC. Prior systemic therapy is defined as any treatment with a chemotherapy agent (or regimen), an immunotherapy agent (or regimen) or an investigational treatment agent (or regimen) against the renal cell carcinoma. Megestrol acetate or medroxyprogesterone will constitute as a prior systemic therapy
* Patients who have at least one uni-dimensional measurable lesion by CT (Computed tomography)-scan or MRI (Magnetic resonance imaging) according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Patients who have an Eastern Co-operative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone marrow, liver , and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening
* Hemoglobin >9.0 g/l
* Absolute neutrophil count ( ANC)>1,500/mm3
* Platelets> or = 100,000/ul
* Total bilirubin < 1.5 x the upper limit of normal
* ALT (Alanine aminotransferase) and AST (Aspartate aminotransferase) < 2.5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer)
* Amylase and lipase < 1.5 x the upper limit of normal
* Serum creatinine < 2.0 x the upper limit of normal
* PT (Prothrombin Time) or INR (International Normalized Ratio) and PTT (Partial Thromboplastin Time) < 1.5 x upper limit of normal (patients who receive anti-coagulation treatment with an agent such as warfarin or heparin will be allowed to participate. For patients on warfarin, close monitoring of at least weekly evaluations will be performed until INR is stable based on a measurement at pre dose, as defined by the local standard of care)

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta [Noninvasive papillary carcinoma], Tis [Carcinoma in situ: "flat tumor"]&T1 [Tumor invades subepithelial connective tissue]) or any cancer curatively treated > 5 years prior to study entry
* Complete renal shut-down requiring hemo- or peritoneal dialysis
* History of cardiac disease : congestive heart failure > NYHA (New York Heart Association) class 2: active cardiovascular disease( MI (Distant metastasis) more than 6 months prior to study entry is allowed); cardiac arrhythmia requiring anti-arrythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension
* Active clinically serious bacterial or fungal infections (>= grade 2 NCI-CTCAE (National Cancer Institute-Common Terminology Criteria for Adverse Events), Version 3)
* Known history of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to this brain tumour site at the time of study entry. Also the patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable provided that the dose is stable for one month prior to and following screening radiographic studies (head CT or MRI at screening always required)
* Patients with seizure disorder requiring medication (such as steroid anti-epileptics)
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Any condition that is unstable or which could jeopardise the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2005-06; Primary Completion 2006-09 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (40):
- United States (9):
  - Sacramento, California
  - Aurora, Colorado
  - Chicago, Illinois
  - Frederick, Maryland
  - Las Vegas, Nevada
  - Cleveland, Ohio
  - Portland, Oregon
  - Dallas, Texas
  - Seattle, Washington
- France (8):
  - Bordeaux
  - Lille
  - Lyon
  - Marseille
  - Nantes
  - Paris
  - Toulouse
  - Villejuif
- Germany (7):
  - Ulm, Baden-Wurttemberg
  - München, Bavaria
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Düsseldorf, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Berlin, State of Berlin
- Poland (6):
  - Gdansk
  - Krakow
  - Poznan
  - Szczecin
  - Warsaw
  - Wroclaw
- Russia (4):
  - Kazan'
  - Kirov
  - Moscow
  - Saint Petersburg
- Ukraine (4):
  - Donetsk
  - Kharkiv
  - Kiev
  - Lviv
- United Kingdom (2):
  - London, London
  - Sutton, Surrey

REFERENCES:
- [Result] Escudier B, Szczylik C, Hutson TE, Demkow T, Staehler M, Rolland F, Negrier S, Laferriere N, Scheuring UJ, Cella D, Shah S, Bukowski RM. Randomized phase II trial of first-line treatment with sorafenib versus interferon Alfa-2a in patients with metastatic renal cell carcinoma. J Clin Oncol. 2009 Mar 10;27(8):1280-9. doi: 10.1200/JCO.2008.19.3342. Epub 2009 Jan 26. PMID 19171708
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The start of enrollment was 14 June 2005 and the last day of enrollment was 12 September 2005.
Pre-assignment Details: All 189 (97 Sorafenib/92 Interferon) randomized subjects were included in the intent to treat (ITT) population, and 187 (97 Sorafenib/90 Interferon) were included in the safety population according to the protocol, which defined eligibility for safety analyses by the prerequisite that a patient had received at least one dose of study medication.
Groups:
- First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg: Subjects received 2 tablets of Sorafenib (200 mg tablets) twice daily (bid) (ie 12-hourly) orally until progression in (= first intervention period, 5.7 months [median] ) and 3 tablets of Sorafenib twice daily (ie 12-hourly) orally until the following progression (= second intervention period, 3.6 months [median]) on a continuous basis.
- First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg: Interferon (IFN) a-2a was administered at a dose of 9 million international units(MIU) subcutaneously three times a week until progression (= first intervention period, 5.6 months [median]). Subjects initially started with a single dose of 3 MIU IFN and increased the dose as rapidly as possible to 9 MIU IFN three times a week within 1 or 2 weeks in first intervention period. After first progression, subjects received 2 tablets of Sorafenib (200 mg tablets) twice daily (BID) (ie 12-hourly) until the next progression (=second intervention period, 5.3 months [median]).
Period: First Intervention (Period 1)
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Started | 97 | 92
Subjects Received Treatment | 97 | 90
Completed | 79 | 67
Not Completed | 18 | 25
Not completed — Adverse Event | 11 | 16
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 4
Not completed — study terminated by the sponsor | 3 | 1
Not completed — protocol driven decision point | 1 | 0
Not completed — investig. decision, not protocol driven | 0 | 1
Not completed — reason not reported | 0 | 1
Period: Second Intervention (Period 2)
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Started | 49 (Not all patients who completed Period 1 (first progression) enter into Period 2) | 61 (Not all patients who completed Period 1 (first progression) enter into Period 2)
Subjects Received Treatment | 49 | 61
Completed | 39 | 39
Not Completed | 10 | 22
Not completed — Adverse Event | 0 | 9
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — study terminated by the sponsor | 2 | 9
Not completed — non compliant with study medication | 1 | 1
Not completed — reason not reported | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg | Total
Number analyzed (Participants) | 97 | 92 | 189
Age, Continuous [Median (Full Range); unit: years] | 62 [34 to 78] | 62.5 [18 to 80] | 62 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 40 | 72
  Male | 65 | 52 | 117
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Category 0 = Fully active, able to carry on all pre-diseases performance without restriction; Category 1 = restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g. light housework, office work).
  participants
    0 | 56 | 49 | 105
    1 | 41 | 43 | 84
Motzer risk factors [Number; unit: participants] — Definition according to Motzer's score (predictive factor): low = no risk factor available; intermediate = 1 or 2 risk factors available; high = 3 or more risk factors available.
  participants
    low | 52 | 47 | 99
    intermediate | 44 | 44 | 88
    high | 1 | 0 | 1
    missing | 0 | 1 | 1
Race [Number; unit: participants]
  White | 68 | 75 | 143
  Asian | 0 | 1 | 1
  Missing | 29 | 16 | 45
Renal Cell Carcinoma (RCC) subtype [Number; unit: participants]
  clear cell | 85 | 81 | 166
  other variant | 12 | 11 | 23
Time since first progression [Median (Full Range); unit: years] | 0.2 [0 to 4.5] | 0.2 [0 to 12.4] | 0.2 [0 to 12.4]
Time since initial diagnosis [Median (Full Range); unit: years] | 0.9 [0.1 to 13.7] | 1 [0.1 to 20.2] | 1 [0.1 to 20.2]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on Independent Radiological Review for the First Intervention Period
Description: Progression-free Survival (PFS) was defined as the time from date of randomization to disease progression (radiological or clinical or death due to any cause, whichever occurs first). Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 97 | 92
months | 5.7 [5.0 to 7.4] | 5.6 [3.7 to 7.4]
Statistical Analysis 1: Comparison: First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg vs First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg; The study was planned to show a 80% improvement in PFS for the group treated with Sorafenib compared to the group treated with Interferon, with a 80% power and a 2-sided type I error of 5%; Test type: Superiority or Other; p = 0.50, Log Rank — The log rank test is stratified by region (western Europe, Eastern Europe, USA) and by Motzer risk category (low, intermediate); Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.61 to 1.27]

2. Secondary Outcome: Progression-free Survival (PFS) Based on Investigator Assessment for the First Intervention Period
Description: as for outcome 1
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 8 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 97 | 92
months | 5.6 [5.4 to 7.5] | 7.0 [5.4 to 8.8]
Statistical Analysis 1: Comparison: First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg vs First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.469, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.882, 95% CI 2-sided [0.628 to 1.239]

3. Secondary Outcome: Disease Control (DC) According to Independent Central Review for the First Intervention Period
Description: Disease Control (DC) was defined as the total number of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD); CR, PR, or SD had to be maintained for at least 28 days from the first demonstration of that rating). CR: disappearance of tumor lesions (TL); PR: a decrease of at least 30% in the sum of TL sizes; SD: steady state of disease; PD: an increase of at least 20% in the sum of TL sizes.
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Measure: Number; unit: participants
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 97 | 92
participants
  disease control (CR or PR or SD) | 77 | 59
  no disease control | 10 | 24
  Unknown | 10 | 9
Statistical Analysis 1: Comparison: First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg vs First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — The Cochran-Mantel-Haenszel statistics was stratified by region and Motzer risk category

4. Secondary Outcome: Disease Control (DC) According to the Investigator Assessment for the First Intervention Period
Description: as for outcome 3
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 8 weeks
Measure: Number; unit: participants
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 97 | 92
participants
  disease control (CR or PR or SD) | 83 | 62
  no disease control | 7 | 24
  Unknown | 7 | 6
Statistical Analysis 1: Comparison: First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg vs First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel — the Cochran-Mantel-Haenszel statistics was stratified by region and Motzer risk category

5. Secondary Outcome: Disease Control (DC) According to the Investigator Assessment for the Second Intervention Period
Description: as for outcome 3
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 8 weeks
Measure: Number; unit: participants
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 49 | 61
participants
  disease control (CR or PR or SD) | 25 | 49
  no disease control | 16 | 6
  Unknown | 8 | 6

6. Secondary Outcome: Analysis of the Quality of Life by Use of the Respiratory Domain of the Functional Assessment of Cancer Therapy-Kidney Symptom Index (FKSI) After Intervention for the First Intervention Period
Description: The FKSI questionnaire comprises 15 questions dispatched within 4 domains (respiratory, pain, general symptoms and overall Quality of Life (QoL)) plus 2 individual items. Each question was answered on a five point scale from 0 (not at all) to 4 (very much) indicating the severity of symptoms. The total score range was from 0 to 60 with higher scores indicating subjects reported fewer kidney cancer related symptoms and concerns. The respiratory domain of the FKSI comprises 2 questions:" I have been short in breath" and "I have been coughing"; its score ranges from 0 to 8.
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: The number of analyzed patients regarding quality of life parameters varied considerably due to missing questionnaires which had not been filled in by patients or invalidity of these questionnaires according to the protocol.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- Sorafenib 400 mg in Period 1: Subjects received 2 tablets of Sorafenib (200 mg tablets) twice daily (bid) (ie 12-hourly) orally until progression in (= first intervention period, 5.7 months [median] ) and 3 tablets of Sorafenib twice daily (ie 12-hourly) orally until the following progression (= second intervention period, 3.6 months [median]) on a continuous basis.
- Interferon Therapy in Period 1: Interferon (IFN) a-2a was administered at a dose of 9 million international units(MIU) subcutaneously three times a week until progression (= first intervention period, 5.6 months [median]). Subjects initially started with a single dose of 3 MIU IFN and increased the dose as rapidly as possible to 9 MIU IFN three times a week within 1 or 2 weeks in first intervention period. After first progression, subjects received 2 tablets of Sorafenib (200 mg tablets) twice daily (BID) (ie 12-hourly) until the next progression (=second intervention period, 5.3 months [median]).
Arm/Group | Sorafenib 400 mg in Period 1 | Interferon Therapy in Period 1
Number analyzed (Participants) | 91 | 87
scores on a scale | 6.4 [3.3 to 9.6] | 5.1 [0.8 to 9.4]
Statistical Analysis 1: Comparison: Sorafenib 400 mg in Period 1 vs Interferon Therapy in Period 1; The least square (LS) means have been adjusted according to the stratification factors (geographical region, Motzer score at baseline) and using the baseline respiratory score as covariate; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis

7. Secondary Outcome: Analysis of the Quality of Life by Use of the Respiratory Domain of the Functional Assessment of Cancer Therapy-Kidney Symptom Index (FKSI) for the Second Intervention Period
Description: as for outcome 6
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- Sorafenib 600 mg (as Dose Escalation After 400 mg): Subjects received 2 tablets of Sorafenib (200 mg tablets) twice daily (bid) (ie 12-hourly) orally until progression in (= first intervention period, 5.7 months [median] ) and 3 tablets of Sorafenib twice daily (ie 12-hourly) orally until the following progression (= second intervention period, 3.6 months [median]) on a continuous basis.
- Sorafenib 400 mg (After Interferon Therapy): Interferon (IFN) a-2a was administered at a dose of 9 million international units(MIU) subcutaneously three times a week until progression (= first intervention period, 5.6 months [median]). Subjects initially started with a single dose of 3 MIU IFN and increased the dose as rapidly as possible to 9 MIU IFN three times a week within 1 or 2 weeks in first intervention period. After first progression, subjects received 2 tablets of Sorafenib (200 mg tablets) twice daily (BID) (ie 12-hourly) until the next progression (=second intervention period, 5.3 months [median]).
Arm/Group | Sorafenib 600 mg (as Dose Escalation After 400 mg) | Sorafenib 400 mg (After Interferon Therapy)
Number analyzed (Participants) | 37 | 42
scores on a scale | 5.7 [-8.2 to 19.7] | 6.4 [-1.2 to 14]

8. Secondary Outcome: Analysis of the Quality of Life by Use of Total Score of the Functional Assessment of Cancer Therapy-Kidney Symptom Index (FKSI) for the First Intervention Period
Description: The FKSI questionnaire comprises 15 questions dispatched within 4 domains (respiratory, pain, general symptoms and overall Quality of Life (QoL)) plus 2 individual items. Each question was answered on a five point scale from 0 (not at all) to 4 (very much) indicating the severity of symptoms. The total score range was from 0 to 60 with higher scores indicating subjects reported fewer kidney cancer related symptoms and concerns.
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib 400 mg in Period 1 | Interferon Therapy in Period 1
Number analyzed (Participants) | 90 | 86
scores on a scale | 40.5 [15.9 to 65.1] | 34.6 [4.4 to 64.8]
Statistical Analysis 1: Comparison: Sorafenib 400 mg in Period 1 vs Interferon Therapy in Period 1; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis

9. Secondary Outcome: Analysis of the Quality of Life by Use of Total Score of the Functional Assessment of Cancer Therapy-Kidney Symptom Index (FKSI) for the Second Intervention Period
Description: as for outcome 8
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib 600 mg (as Dose Escalation After 400 mg) | Sorafenib 400 mg (After Interferon Therapy)
Number analyzed (Participants) | 37 | 42
scores on a scale | 34.6 [6.3 to 62.9] | 42.3 [9.5 to 75.2]

10. Secondary Outcome: Analysis of the Quality of Life (QoL) by Use of Functional Assessment of Cancer Therapy-Biologic-response Modifiers (FACT-BRM) for the First Intervention Period
Description: The FACT-BRM comprises 40 questions within 6 domains (physical well being, social/family well being, emotional well being, additional concern: physical, and additional concern: emotional). Each question was answered on a five point scale from 0 (not at all) to 4 (very much). The total score range is from 0 to 160 with higher scores indicating better QoL.
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib 400 mg in Period 1 | Interferon Therapy in Period 1
Number analyzed (Participants) | 89 | 86
scores on a scale | 104 [29 to 179] | 93 [-9 to 195]
Statistical Analysis 1: Comparison: Sorafenib 400 mg in Period 1 vs Interferon Therapy in Period 1; The least square (LS) means have been adjusted according to the stratification factors (geographical region, Motzer score at baseline); Test type: Superiority or Other; p = 0.073, Mixed Models Analysis

11. Secondary Outcome: Analysis of the Quality of Life (QoL) by Use of Functional Assessment of Cancer Therapy-Biologic-response Modifiers (FACT-BRM) for the Second Intervention Period
Description: as for outcome 10
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib 600 mg (as Dose Escalation After 400 mg) | Sorafenib 400 mg (After Interferon Therapy)
Number analyzed (Participants) | 37 | 40
scores on a scale | 89.7 [18.2 to 161.1] | 108.4 [17.6 to 199.2]

12. Secondary Outcome: Analysis of the Treatment Tolerability (Effectiveness) by Use of Treatment Satisfaction Questionnaire for Medication (TSQM) for the First Intervention Period
Description: The TSQM comprises 14 questions dispatched within 4 domains (effectiveness, side effects, convenience, and global satisfaction). Each question was answered on either a 5-point or 7-point scale. Each domain score can vary from 0 to 100 with higher scores indicating subject reported higher effectiveness of treatment, less bothered by side-effects, more convenient use of medication and overall greater satisfaction with the treatment. No total score is calculated.
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib 400 mg in Period 1 | Interferon Therapy in Period 1
Number analyzed (Participants) | 29 | 34
scores on a scale | 52 [44 to 61] | 42 [34 to 50]
Statistical Analysis 1: Comparison: Sorafenib 400 mg in Period 1 vs Interferon Therapy in Period 1; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.067, Mixed Models Analysis

13. Secondary Outcome: Analysis of the Treatment Tolerability (Side Effects) by Use of Treatment Satisfaction Questionnaire for Medication (TSQM) for the First Intervention Period
Description: as for outcome 12
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib 400 mg in Period 1 | Interferon Therapy in Period 1
Number analyzed (Participants) | 27 | 30
scores on a scale | 63 [54 to 72] | 46 [37 to 54]
Statistical Analysis 1: Comparison: Sorafenib 400 mg in Period 1 vs Interferon Therapy in Period 1; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis

14. Secondary Outcome: Analysis of the Treatment Tolerability (Convenience) by Use of Treatment Satisfaction Questionnaire for Medication (TSQM) for the First Intervention Period
Description: as for outcome 12
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib 400 mg in Period 1 | Interferon Therapy in Period 1
Number analyzed (Participants) | 30 | 33
scores on a scale | 82 [75 to 89] | 66 [60 to 73]
Statistical Analysis 1: Comparison: Sorafenib 400 mg in Period 1 vs Interferon Therapy in Period 1; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis

15. Secondary Outcome: Analysis of the Treatment Tolerability (Global Satisfaction) by Use of Treatment Satisfaction Questionnaire for Medication (TSQM) for the First Intervention Period
Description: as for outcome 12
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib 400 mg in Period 1 | Interferon Therapy in Period 1
Number analyzed (Participants) | 30 | 33
scores on a scale | 60 [51 to 70] | 46 [37 to 55]
Statistical Analysis 1: Comparison: Sorafenib 400 mg in Period 1 vs Interferon Therapy in Period 1; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis

16. Secondary Outcome: Analysis of the Treatment Tolerability (Effectiveness) by Use of Treatment Satisfaction Questionnaire for Medication (TSQM) for the Second Intervention Period
Description: as for outcome 12
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib 600 mg (as Dose Escalation After 400 mg) | Sorafenib 400 mg (After Interferon Therapy)
Number analyzed (Participants) | 10 | 9
scores on a scale | 56.9 [40.6 to 73.1] | 40.3 [22.1 to 58.5]

17. Secondary Outcome: Analysis of the Treatment Tolerability (Side Effects) by Use of Treatment Satisfaction Questionnaire for Medication (TSQM) for the Second Intervention Period
Description: as for outcome 12
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib 600 mg (as Dose Escalation After 400 mg) | Sorafenib 400 mg (After Interferon Therapy)
Number analyzed (Participants) | 10 | 8
scores on a scale | 61.3 [43.2 to 79.3] | 57.6 [37.4 to 77.8]

18. Secondary Outcome: Analysis of the Treatment Tolerability (Convenience) by Use of Treatment Satisfaction Questionnaire for Medication (TSQM) for the Second Intervention Period
Description: as for outcome 12
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib 600 mg (as Dose Escalation After 400 mg) | Sorafenib 400 mg (After Interferon Therapy)
Number analyzed (Participants) | 11 | 9
scores on a scale | 86.5 [74.7 to 98.3] | 82.5 [68.9 to 96.1]

19. Secondary Outcome: Analysis of the Treatment Tolerability (Global Satisfaction) by Use of Treatment Satisfaction Questionnaire for Medication (TSQM) for the Second Intervention Period
Description: as for outcome 12
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib 600 mg (as Dose Escalation After 400 mg) | Sorafenib 400 mg (After Interferon Therapy)
Number analyzed (Participants) | 11 | 8
scores on a scale | 39.9 [17.1 to 62.7] | 35.4 [9.4 to 61.8]

20. Secondary Outcome: Tumor Response According to the Independent Radiological Review for the First Intervention Period
Description: Tumor Response (= Best Overall Response) of a subject was defined as the best tumor response (confirmed Complete Response (CR), confirmed Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD)) observed during trial period assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. CR was defined as disappearance of tumor lesions, PR was defined as a decrease of at least 30% in the sum of tumor lesion sizes, SD was defined as steady state of disease, PD was defined as an increase of at least 20% in the sum of tumor lesions sizes.
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Measure: Number; unit: participants
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 97 | 92
participants
  Complete Response (CR) | 0 | 1
  Partial Response (PR) | 5 | 7
  Stable Disease (SD) | 72 | 51
  Progressive Disease (PD) | 10 | 24
  Not Evaluated | 10 | 9

21. Secondary Outcome: Tumor Response According to the Investigator Assessment for the First Intervention Period
Description: as for outcome 20
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 8 weeks
Measure: Number; unit: participants
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 97 | 92
participants
  Complete Response (CR) | 0 | 1
  Partial Response (PR) | 21 | 13
  Stable Disease (SD) | 62 | 48
  Progressive Disease (PD) | 7 | 24
  Not Evaluated | 7 | 6

22. Secondary Outcome: Tumor Response According to the Investigator Assessment for the Second Intervention Period
Description: as for outcome 20
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 8 weeks
Measure: Number; unit: participants
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 49 | 61
participants
  Complete Response (CR) | 0 | 1
  Partial Response (PR) | 0 | 11
  Stable Disease (SD) | 25 | 37
  Progressive Disease (PD) | 16 | 6
  Not Evaluated | 8 | 6

23. Secondary Outcome: Progression Free Survival According to the Investigator Assessment (Second Intervention Period)
Description: as for outcome 1
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 8 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 49 | 61
months | 4.5 [2.4 to 6.5] | 5.5 [3.8 to 7.1]

24. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 8 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 97 | 92
months | 14.8 [11.3 to 17.7] | 26.9 [18.3 to 33.8]
Statistical Analysis 1: Comparison: First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg vs First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg; Test type: Superiority or Other; p = 0.014, Log Rank

25. Secondary Outcome: Slope - Change in Trough Concentration/Cycle
Description: Plasma samples were collected prior to dosing every 4 weeks after the patient reached steady-state (at least 10 days at 400 mg BID (bis in die, twice daily)) to assess any potential trends in trough concentration over time.
Time Frame: From start of treatment of the first subject until 15 months later assessed every 4 weeks.
Population: Patients who started on Sorafenib, not Interferon, and had been at the same dose (400 mg) for at least 10 days were considered valid for the analysis. Concentrations collected between 10-14 hours from the last dose were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: 100*(mg/L/cycle)
Groups:
- First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600mg: Subjects received 2 tablets of Sorafenib (200 mg tablets) twice daily (bid) (ie 12-hourly) orally until progression in (= first intervention period, 5.7 months [median] ) and 3 tablets of Sorafenib twice daily (ie 12-hourly) orally until the following progression (= second intervention period, 3.6 months [median]) on a continuous basis.
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600mg
Number analyzed (Participants) | 24
100*(mg/L/cycle) | -8.3 [-29.6 to 12.9]

26. Secondary Outcome: Average of All Trough Plasma Concentrations
Description: Plasma samples were collected prior to dosing every 4 weeks after the patient reached steady-state (at least 10 days at 400 mg BID).
Time Frame: From start of treatment of the first subject until 15 months later assessed every 4 weeks.
Population: Patients who started on Sorafenib, not Interferon, and had been at the same dose (400 mg or 600 mg BID) for at least 10 days were considered valid for the analysis. Concentrations collected between 10-14 hours from the last dose were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: 100*mg/L
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600mg
Number analyzed (Participants) | 24
100*mg/L | 93.9 [77.1 to 114.3]

27. Secondary Outcome: Duration of Response According to the Independent Radiological Review for the First Intervention Period
Description: Duration of Response was defined as the time from date of first response (Complete Response (CR) or Partial Response (PR)) to the date when Progressive Disease (PD) is first documented or to the date of death, whichever occurs first. Subjects still having CR or PR at the time of analysis were censored at their last date of last contact
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Measure: Median (Full Range); unit: months
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 5 | 8
months | 7.5 [7.5 to 7.5] | 7.7 [2.1 to 7.8]

28. Secondary Outcome: Duration of Response According to the Investigator Assessment for the First Intervention Period
Description: as for outcome 27
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 8 weeks
Measure: Median (Full Range); unit: months
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 21 | 14
months | 4.4 [1.2 to 22] | 9.2 [1.5 to 19.7]

29. Secondary Outcome: Duration of Response According to the Investigator Assessment for the Second Intervention Period
Description: as for outcome 27
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 8 weeks
Measure: Median (Full Range); unit: months
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 0 | 12
months |  | 5.5 [1.1 to 16.7]

30. Secondary Outcome: Time to Response According to the Independent Radiological Review for the First Intervention Period
Description: Time to Response (TTR) for subjects who achieved a response (Complete Response (CR) or Partial Response (PR) with confirmation was defined as the time from date of randomization to the earliest date that the response was first documented
Time Frame: From randomization of the first subject until 15 months later, assessed every 8 weeks
Measure: Median (Full Range); unit: months
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 5 | 8
months | 1.8 [1.7 to 3.7] | 5.4 [3.7 to 11]

31. Secondary Outcome: Time to Response According to the Investigator Assessment for the First Intervention Period
Description: as for outcome 30
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 4 weeks
Measure: Median (Full Range); unit: months
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 21 | 14
months | 3.5 [1.6 to 11.1] | 5.4 [1.2 to 18.3]

32. Secondary Outcome: Time to Response According to the Investigator Assessment for the Second Intervention Period
Description: Time to Response (TTR) for subjects who achieved a response (Complete Response (CR) or Partial Response (PR) with confirmation) was defined as the time from date of randomization to the earliest date that the response was first documented
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 4 weeks
Measure: Median (Full Range); unit: months
Arm/Group | First Sorafenib (Nexavar, BAY43-9006) 400 mg Then 600 mg | First Interferon Then Sorafenib (Nexavar, BAY43-9006) 400 mg
Number analyzed (Participants) | 0 | 12
months |  | 1.7 [1.6 to 5.4]

33. Secondary Outcome: Analysis of the Eastern Co-operative Oncology Group (ECOG) Status at the End of the First Intervention Period
Description: Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale that measures how cancer affects the daily life of a patient on an ordinal scale from grade 0 (best) to grade 5 (worst).
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 4 weeks
Population: At the time of the analysis, only 95 subjects in Sorafenib 400 mg bid group and 89 in Interferon group were documented by study investigators due to various reasons (drop-out of patients by AEs, death etc.)
Measure: Number; unit: participants
Arm/Group | Sorafenib 400 mg in Period 1 | Interferon Therapy in Period 1
Number analyzed (Participants) | 95 | 89
participants
  0= Fully active without restriction | 20 | 19
  1= Restricted in physically strenuous activity | 48 | 42
  2= Ambulatory, capable of all selfcare | 20 | 21
  3= Capable of limited selfcare | 5 | 5
  4= Completely disabled | 1 | 2
  5= Dead | 1 | 0

34. Secondary Outcome: Analysis of the Eastern Co-operative Oncology Group (ECOG) Status at the End of the Second Intervention Period
Description: as for outcome 33
Time Frame: From randomization of the first subject until 3 years and 9 months later, assessed every 4 weeks
Population: At the time of the analysis, only 45 subjects in Sorafenib 400/600 mg bid group and 58 in Interferon/Sorafenib 400 mg bid group were documented by study investigators due to various reasons (drop-out of patients by AEs, death etc.)
Measure: Number; unit: participant s
Arm/Group | Sorafenib 600 mg (as Dose Escalation After 400 mg) | Sorafenib 400 mg (After Interferon Therapy)
Number analyzed (Participants) | 45 | 58
participant s
  0= Fully active without restriction | 5 | 16
  1= Restricted in physically strenuous activity | 25 | 26
  2= Ambulatory, capable of all selfcare | 10 | 10
  3= Capable of limited selfcare | 4 | 5
  4= Completely disabled | 1 | 1
  5= Dead | 0 | 0

ADVERSE EVENTS:
Description: Acronyms and abbreviations used: Common Terminology Criteria for Adverse Events (CTCAE); Not Otherwise Specified (NOS); Gastrointestinal (GI); Absolute Neutrophil Count (ANC); Alanine aminotransferase (ALT); Aspartate aminotransferase (AST); Central nervous system (CNS); Acute respiratory distress syndrome (ARDS)
Arm/Group | Sorafenib 400 mg in Period 1 | Interferon Therapy in Period 1 | Sorafenib 600 mg (as Dose Escalation After 400 mg) | Sorafenib 400 mg (After Interferon Therapy)
Serious Adverse Events (participants affected / at risk) | 47/97 | 36/90 | 14/49 | 30/61
Other Adverse Events (participants affected / at risk) | 93/97 | 84/90 | 40/49 | 55/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib 400 mg in Period 1 (N=97) | Interferon Therapy in Period 1 (N=90) | Sorafenib 600 mg (as Dose Escalation After 400 mg) (N=49) | Sorafenib 400 mg (After Interferon Therapy) (N=61)
allergic reaction (Immune system disorders) | 1 | 1 | 0 | 0
auditory / ear - other (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
hemoglobin (Blood and lymphatic system disorders) | 2 | 6 | 2 | 4
platelets (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
conduction abnormality, asystole (Cardiac disorders) | 0 | 1 | 0 | 0
supraventricular arrhythmia, supraventricular arrhythmi (Cardiac disorders) | 0 | 1 | 0 | 0
supraventricular arrhythmia, atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
cardiopulmonary arrest (Cardiac disorders) | 1 | 0 | 0 | 0
cardiac ischemia / infarction (Cardiac disorders) | 1 | 1 | 0 | 1
cardiac general - other (Cardiac disorders) | 1 | 2 | 1 | 4
death not associated with CTCAE term, death NOS (General disorders) | 1 | 0 | 0 | 0
death not associated with CTCAE term, disease progress (General disorders) | 10 | 1 | 2 | 7
fever (General disorders) | 1 | 0 | 0 | 0
fatigue (General disorders) | 1 | 3 | 0 | 2
constitutional symptoms - other (General disorders) | 6 | 4 | 0 | 5
ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1
constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
dehydration (Gastrointestinal disorders) | 0 | 1 | 0 | 1
diarrhea (Gastrointestinal disorders) | 2 | 0 | 0 | 2
nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 1
obstruction, GI, stomach (Gastrointestinal disorders) | 1 | 0 | 0 | 0
perforation, GI, colon (Gastrointestinal disorders) | 0 | 1 | 0 | 0
vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 1
ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GI - other (Gastrointestinal disorders) | 0 | 0 | 0 | 1
hematoma (Vascular disorders) | 0 | 1 | 0 | 0
hemorrhage, GI, colon (Vascular disorders) | 0 | 1 | 0 | 0
hemorrhage, GI, stomach (Vascular disorders) | 0 | 1 | 0 | 0
hemorrhage, GI, lower GI NOS (Vascular disorders) | 0 | 1 | 0 | 1
hemorrhage, GI, upper GI NOS (Vascular disorders) | 0 | 2 | 0 | 0
hemorrhage - other (Vascular disorders) | 2 | 0 | 0 | 0
hemorrhage pulmonary, bronchopulmonary NOS (Vascular disorders) | 1 | 0 | 1 | 0
hemorrhage, GI, anus (Vascular disorders) | 0 | 0 | 1 | 0
hemorrhage, GI, varices (rectal) (Vascular disorders) | 0 | 0 | 1 | 0
hepatobiliary - other (Hepatobiliary disorders) | 0 | 1 | 0 | 0
liver dysfunction (Hepatobiliary disorders) | 0 | 0 | 0 | 1
infection (documented clinically), appendix (Infections and infestations) | 0 | 1 | 0 | 0
infection with normal ANC, abdomen NOS (Infections and infestations) | 1 | 0 | 0 | 0
infection with normal ANC, lung (pneumonia) (Infections and infestations) | 1 | 1 | 0 | 0
infection with unknown ANC, bronchus (Infections and infestations) | 1 | 0 | 0 | 0
infection with unknown ANC, upper airway NOS (Infections and infestations) | 1 | 0 | 0 | 0
infection (documented clinically), lung (pneumonia) (Infections and infestations) | 0 | 0 | 1 | 0
infection - other (Infections and infestations) | 0 | 0 | 0 | 3
fracture (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0
edema: limb (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
ALT (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
AST (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
metabolic / lab - other (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
CNS ischemia (Nervous system disorders) | 1 | 1 | 0 | 0
confusion (Nervous system disorders) | 0 | 3 | 0 | 0
dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0
mood alteration, depression (Nervous system disorders) | 0 | 1 | 0 | 0
neurology - other (Nervous system disorders) | 1 | 1 | 0 | 3
seizure (Nervous system disorders) | 2 | 0 | 0 | 0
somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
speech impairment (Nervous system disorders) | 0 | 0 | 0 | 1
pain, back (General disorders) | 1 | 0 | 0 | 0
pain, chest / thorax NOS (General disorders) | 1 | 0 | 0 | 1
pain, extremity - limb (General disorders) | 0 | 1 | 1 | 1
pain, tumor pain (General disorders) | 1 | 0 | 1 | 0
pain, abdomen NOS (General disorders) | 3 | 1 | 0 | 1
pain, head / headache (General disorders) | 1 | 0 | 0 | 0
pain, bone (General disorders) | 2 | 0 | 1 | 0
pain, other (General disorders) | 1 | 0 | 1 | 1
pain, joint (General disorders) | 0 | 0 | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
airway obstruction, bronchus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
renal failure (Renal and urinary disorders) | 3 | 0 | 0 | 0
urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
secondary malignancy (possibly related to cancer treat) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
thrombosis / thrombus / embolism (Vascular disorders) | 2 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib 400 mg in Period 1 (N=97) | Interferon Therapy in Period 1 (N=90) | Sorafenib 600 mg (as Dose Escalation After 400 mg) (N=49) | Sorafenib 400 mg (After Interferon Therapy) (N=61)
rhinitis (Immune system disorders) | 6 | 1 | 0 | 0
neutrophils (Blood and lymphatic system disorders) | 2 | 13 | 0 | 0
hemoglobin (Blood and lymphatic system disorders) | 14 | 23 | 10 | 8
platelets (Blood and lymphatic system disorders) | 1 | 11 | 2 | 4
leukocytes (Blood and lymphatic system disorders) | 2 | 11 | 0 | 0
lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 3
hypertension (Cardiac disorders) | 24 | 7 | 1 | 13
fever (General disorders) | 10 | 30 | 2 | 4
insomnia (General disorders) | 2 | 8 | 0 | 0
fatigue (General disorders) | 48 | 41 | 16 | 22
weight loss (General disorders) | 26 | 24 | 12 | 10
constitutional symptoms - other (General disorders) | 7 | 11 | 3 | 4
rigors / chills (General disorders) | 1 | 10 | 0 | 0
anorexia (Gastrointestinal disorders) | 34 | 28 | 11 | 8
constipation (Gastrointestinal disorders) | 12 | 2 | 3 | 9
diarrhea (Gastrointestinal disorders) | 54 | 14 | 12 | 31
dry mouth (Gastrointestinal disorders) | 5 | 1 | 0 | 0
mucositis (functional / symptomatic), oral cavity (Gastrointestinal disorders) | 12 | 2 | 1 | 8
mucositis (clinical exam), oral cavity (Gastrointestinal disorders) | 5 | 1 | 0 | 4
nausea (Gastrointestinal disorders) | 24 | 26 | 5 | 14
taste alteration (Gastrointestinal disorders) | 6 | 6 | 0 | 0
vomiting (Gastrointestinal disorders) | 18 | 15 | 5 | 9
hemorrhage pulmonary, nose (Vascular disorders) | 5 | 1 | 0 | 0
infection with normal ANC, urinary tract NOS (Infections and infestations) | 7 | 2 | 3 | 0
infection - other (Infections and infestations) | 12 | 2 | 5 | 7
infection with unknown ANC, urinary tract NOS (Infections and infestations) | 5 | 2 | 0 | 0
infection (documented clinically), urinary tract NOS (Infections and infestations) | 0 | 0 | 0 | 4
infection with normal ANC, upper airway NOS (Infections and infestations) | 0 | 0 | 3 | 1
edema: limb (Blood and lymphatic system disorders) | 4 | 5 | 5 | 2
ALT (Metabolism and nutrition disorders) | 5 | 8 | 0 | 0
AST (Metabolism and nutrition disorders) | 6 | 9 | 0 | 0
creatinine (Metabolism and nutrition disorders) | 3 | 6 | 3 | 0
hyperuricemia (Metabolism and nutrition disorders) | 8 | 2 | 5 | 5
lipase (Metabolism and nutrition disorders) | 16 | 5 | 1 | 7
amylase (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3
hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4
hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 2
hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 4
hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1
metabolic / lab - other (Metabolism and nutrition disorders) | 0 | 0 | 3 | 4
confusion (Nervous system disorders) | 5 | 4 | 0 | 0
dizziness (Nervous system disorders) | 5 | 9 | 0 | 0
mood alteration, depression (Nervous system disorders) | 5 | 15 | 4 | 3
neuropathy: sensory (Nervous system disorders) | 6 | 1 | 3 | 4
pain, back (General disorders) | 12 | 5 | 2 | 4
pain, extremity - limb (General disorders) | 7 | 7 | 1 | 7
pain, tumor pain (General disorders) | 4 | 5 | 0 | 0
pain, abdomen NOS (General disorders) | 14 | 10 | 3 | 7
pain, head / headache (General disorders) | 5 | 13 | 0 | 5
pain, joint (General disorders) | 4 | 5 | 3 | 3
pain, muscle (General disorders) | 9 | 6 | 0 | 4
pain, bone (General disorders) | 9 | 8 | 4 | 1
pain, other (General disorders) | 18 | 10 | 5 | 9
pain, neuralgia / peripheral nerve (General disorders) | 5 | 1 | 0 | 0
pain, stomach (General disorders) | 5 | 4 | 0 | 0
pain, chest / thorax NOS (General disorders) | 0 | 0 | 1 | 5
cough (Respiratory, thoracic and mediastinal disorders) | 12 | 15 | 3 | 6
dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 13 | 10 | 4 | 4
voice changes (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 0 | 0
renal - other (Renal and urinary disorders) | 6 | 0 | 0 | 0
alopecia (Skin and subcutaneous tissue disorders) | 40 | 6 | 2 | 17
dry skin (Skin and subcutaneous tissue disorders) | 10 | 9 | 2 | 6
hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 57 | 4 | 8 | 28
dermatology - other (Skin and subcutaneous tissue disorders) | 7 | 2 | 4 | 5
pruritus (Skin and subcutaneous tissue disorders) | 14 | 12 | 1 | 6
rash / desquamation (Skin and subcutaneous tissue disorders) | 40 | 8 | 4 | 17
flu-like syndrome (General disorders) | 5 | 20 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication will be discussed with the sponsor prior to release and written consent of the sponsor will be obtained. A draft manuscript of the publication or abstract must be sent to sponsor thirty days in advance of submission.